CLINICAL TRIAL: NCT00156429
Title: Genetic Predictors of Outcome in HCM Patients
Status: Terminated | Type: Observational
Why Stopped: Preliminary analyses did not reveal significant associations.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Timothy Wong, Assistant Professor, University of Pittsburgh
Other Study IDs: 0507025; 0507025
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: genetic testing
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for DNA analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective review of the data available on patients and their family members with HCM and prospective follow-up of this cohort for clinical outcome and diagnostic studies. Genetic samples are being examined in this cohort to determine whether certain to determine whether certain beta-AR polymorphisms as well as other common genetic polymorphisms are associated with different morphological features, such as LVH in patients with HCM and whether these polymorphisms influence the clinical course and outcome in patients with HCM. For that purpose, we will build a database with clinical information including serial echocardiographic measurements for patients with HCM that have regular follow up and test them for beta-AR polymorphisms as well as other common genetic polymorphisms and other known cardiac-related polymorphisms that can potentially contribute to the morphologic differences seen in patients with HCM.

DETAILED DESCRIPTION:
This is a retrospective review of the data available on patients and their family members with HCM and prospective follow-up of this cohort for clinical outcome and diagnostic studies. Genetic samples are being examined in this cohort to determine whether certain to determine whether certain beta-AR polymorphisms as well as other common genetic polymorphisms are associated with different morphological features, such as LVH in patients with HCM and whether these polymorphisms influence the clinical course and outcome in patients with HCM. For that purpose, we will build a database with clinical information including serial echocardiographic measurements for patients with HCM that have regular follow up and test them for beta-AR polymorphisms as well as other common genetic polymorphisms and other known cardiac-related polymorphisms that can potentially contribute to the morphologic differences seen in patients with HCM.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Diagnosed with HCM defined by the presence of left ventricular hypertrophy with minimal wall thickness >/= 15mm without the presence of hypertension or systemic disease that can account for the degree of hypertrophy.

Exclusion Criteria:

* Hypertension present prior to the diagnosis of HCM
* aortic stenosis with aortic valve area < 1cm2
* known systemic disease that can cause LVH, such as infiltrative diseases
* able and willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HCM
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-04-22 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Genetic testing | Day 1 at the time of enrollment
  AR polymorphisms will be correlated to progression of LVH and clinical outcome in patients with HCM.

CONTACTS AND LOCATIONS:
Overall Officials: Samir F. Saba, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States